CLINICAL TRIAL: NCT04810169
Title: Towards Participatory Paediatric Asthma Action Plans
Acronym: PACAP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200937; 2020-A02722-37 (Other: ID-RCB)
Record Dates: First submitted 2021-03-08; First posted 2021-03-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: Action plan; Asthma; Paediatric
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smart inhaler: Children with smart inhaler
  Interventions: Device: Smart inhaler

INTERVENTIONS:
Device: Smart inhaler — * Automatic record (number of actuations and their timing) of the use of the emergency treatment through the smart inhaler
  * Questionnaire sent to the parents at each use of the smart inhaler to get information regarding the reason of use and the efficacy of the treatment given

SUMMARY:
Asthma is the most common chronic disease in children. The management of asthma attacks at home is based on asthma action plans that are very heterogeneous and reflect the diversity of recommendations on this subject. The purpose of this study is to observe using smartinhalers how children and their families use their emergency treatment at home in case of asthma symptoms and asthma attacks, to allow building new recommendations based not only on the literature, but also on real-world data.

DETAILED DESCRIPTION:
Asthma is the most common chronic disease in children. Asthma exacerbations are responsible for many unscheduled consultations by paediatricians and general practitioners, numerous emergency room visits and frequent hospitalizations

Asthma action plans are documents given to families and schools to give the actions to be taken in the event of an asthma attack occurring in the family or school environment. They are recommended by all learned societies, because, combined with patient education and regular consultations, they reduce the need for unscheduled care.

The main drug in the action plan is the emergency treatment, i.e. a short-acting bronchodilator (SABA). However, the doses of SABA to be used vary widely depending on the recommendations. For children up to 5 years of age, the international board of the Global Initiative for Asthma (GINA) suggests limiting the home dose to 2 puffs of 100μg every 20 minutes, to be repeated twice before consulting a physician if there is no improvement. This dose is increased to 4-10 puffs every 20 minutes in children 6 years and older. The British Thoracic Society in the United Kingdom advises administering salbutamol puffs one at a time, 30 to 60 seconds apart, until symptoms improve, with a maximum of 10 puffs. In France, the Groupe de Recherche sur les Avancées en PneumoPédiatrie (GRAPP) recommends to administer higher doses of salbutamol at home, up to one puff per 2 kg of weight, with a maximum of 10 to 15 puffs, to be repeated every 20 minutes for one hour, before giving oral corticosteroids. These very heterogeneous protocols reflect the diversity of doses proposed in the literature, and the paucity of clinical research data that makes it impossible to determine whether one approach is better than another. A study that looked at the goals of parents of children with asthma highlighted that this heterogeneity of practices is a source of stress for families: "I would like one plan and not ten" explained one parent; "I would like a plan that doesn't change all the time" reported another.

Harmonization of practices is necessary in order to provide families and school physicians nurses with a consistent approach..

The aim of this study is therefore to observe, using inhalers connected to salbutamol inhalers (smart inhalers), how families manage an asthma exacerbation at home, and to integrate these data into the establishment of future recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Parent of 18 years or more
* Parent with a smartphone compatible with a smart inhaler
* Parent with child who :

  * is 3 years to 11 years 11 months old
  * has physician-diagnosed asthma diagnosis
  * has a prescription of emergency treatment in case of asthma symptom
* Non-opposition of the legal guardian

Exclusion Criteria:

* Refuse to participate at the study
* Difficulty reading and/or understanding French language
* Technical problem (malfunction) with the smart inhalers and/or the associated mobile application during the initial test with the parent's smartphone

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with asthma
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Mean number of emergency-treatments administered in the first two hours of management | 6 months
  Mean number of emergency-treatments administered in the first two hours of management, depending on the symptoms initially presented by the child (cough, wheezing, dyspnea, or respiratory distress) or an association of symptoms, which led to the disappearance of the symptom(s) that prompted the initiation of salbutamol.

SECONDARY OUTCOMES:
Improvement of one or more symptoms | 6 months
  Improvement of the symptom(s), defined in a binary manner as an improvement reported by parents on the mobile application within 24 hours of the onset of the symptom(s).
Elimination of one or more symptoms | 6 months
  Elimination of one or more symptoms defined in a binary manner (success/failure) by not using salbutamol for an asthmatic symptom within 24 hours of the onset of the symptom or symptoms.
Compliance score for action plan | 6 months
  taking into account the number of salbutamol puffs administered compared to the recommended number of salbutamol puffs, the duration between salbutamol puffs compared to the recommended duration, and the sequence of actions performed (including corticosteroids and use of the healthcare system) compared to the recommended sequence of actions - This score will be calculated as follows: (Number of expected actions on the action plan and according to the evolution of symptoms - Number of actions recorded by the smartinhalers and on the research application) / number of expected actions * 100.
Overtreatment by families | 6 months
  Family overuse of salbutamol, defined as ((number of puffs recorded - number of puffs expected)/(number of puffs expected) * 100) strictly greater than 50%.
Undertreatment by families | 6 months
  Under-use of salbutamol by families, defined as ((number of puffs recorded - number of puffs expected)/(number of puffs expected) * 100) strictly less than -50%.

CONTACTS AND LOCATIONS:
Overall Officials: David DRUMMOND, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marguet C, Michelet I, Couderc L, Lubrano M. [Management of acute asthma exacerbation in childhood: French recommendations]. Arch Pediatr. 2009 Jun;16(6):505-7. doi: 10.1016/S0929-693X(09)74046-1. No abstract available. French. PMID 19541064
- [Background] Pinnock H, Parke HL, Panagioti M, Daines L, Pearce G, Epiphaniou E, Bower P, Sheikh A, Griffiths CJ, Taylor SJ; PRISMS and RECURSIVE groups. Systematic meta-review of supported self-management for asthma: a healthcare perspective. BMC Med. 2017 Mar 17;15(1):64. doi: 10.1186/s12916-017-0823-7. PMID 28302126
- [Background] Heidi M, Emily K, Benjamin H, Michael C, Robert K, Mitch B, Chris G, Mando W, Andrew B. Patient reported outcomes for preschool children with recurrent wheeze. NPJ Prim Care Respir Med. 2019 Mar 26;29(1):7. doi: 10.1038/s41533-019-0120-3. PMID 30914646
- [Result] Gonsard A, Giovannini-Chami L, Cros P, Masson A, Menetrey C, Mordacq C, Cisterne C, Personnic J, Roy C, Poirault C, Abou Taam R, Hadchouel A, Pirojoc A, Delacourt C, Drummond D. Home use of short-acting beta agonists by children with asthma: a multicentre digital prospective study. Arch Dis Child. 2025 Aug 18;110(9):701-705. doi: 10.1136/archdischild-2024-327447. PMID 40169179
- See also: Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention. (2020) — https://ginasthma.org/gina-reports/